CLINICAL TRIAL: NCT06899334
Title: Direct Comparison of Altered States of Consciousness Induced by LSD, Psilocybin, and DMT in a Randomized, Placebo-controlled, Cross-over Trial in Healthy Participants (LPD-Study)
Brief Title: Direct Comparison of Altered States of Consciousness Induced by LSD, Psilocybin, and DMT in Healthy Participants
Acronym: LPD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BASEC 2024-01445
Record Dates: First submitted 2025-03-14; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: Psychedelics; LSD; Psilocybin; DMT
MeSH Terms: interventions — Lysergic Acid Diethylamide; Psilocybin

STUDY DESIGN:
Intervention Model Description: 4-period, random order, placebo-controlled, double-blind cross-over study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LSD (Experimental): 150 µg lysergic acid diethylamide followed by 20 mg ketanserin intravenously after 3 h
  Interventions: Drug: LSD
- Psilocybin (Experimental): 30 mg Psilocybin followed by 20 mg ketanserin intravenously after 3 h
  Interventions: Drug: Psilocybin
- DMT (Experimental): Dose escalating DMT intravenous infusion up to 2 mg/min followed by 20 mg ketanserin intravenously after 3 h
  Interventions: Drug: DMT
- Placebo (Placebo Comparator): Placebo followed by 20 mg ketanserin intravenously after 3 h
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LSD — A moderate to high oral dose of 150 µg LSD will be administered followed by 20 mg intravenous ketanserin after 3 h
  Arms: LSD
Drug: Psilocybin — A moderate to high oral dose of 30 mg psilocybin will be administered followed by 20 mg intravenous ketanserin after 3 h
  Arms: Psilocybin
Drug: DMT — A moderate to high, dose-escalating, intravenous infusion up to 2 mg/min DMT will be administered followed by 20 mg intravenous ketanserin after 3 h
  Arms: DMT
Drug: Placebo — An oral and an intravenous placebo will be administered followed by 20 mg intravenous ketanserin after 3 h
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine whether equivalent moderately high doses of LSD, psilocybin, and DMT produce qualitatively similar peak effects when the effect duration is standardized with ketanserin. A DMT infusion mimicking oral LSD and psilocybin administrations will be tested, as well as intravenously administered ketanserin.

DETAILED DESCRIPTION:
Lysergic acid diethylamide (LSD), psilocybin, and N,N-dimethyltryptamine (DMT) are serotonergic hallucinogens (psychedelics) and currently investigated as therapeutic tools for the treatment of various psychiatric disorders. They are usually administered in a dose range which induces an alteration of consciousness via the stimulation of the serotonin (5-HT)2A receptor. However, there are differences in the receptor activation profiles between the three substances that may induce different subjective effects. Moreover, they exhibit different pharmacokinetic qualities. In comparative studies of LSD and psilocybin blinding was impaired by the different duration of subjective effects. This study aims to ensure blinding by ending all experiences at the same time with the 5HT2A antagonist ketanserin. Moreover, no study has yet directly compared DMT to LSD and psilocybin. The DMT infusion will be modeled in accordance with the course of an oral LSD and psilocybin administration. Therefore, the LPD-study compares the acute and subacute effects of LSD, psilocybin, and DMT while standardizing the time course and the duration of action for all substances.

ELIGIBILITY:
Inclusion Criteria:

1. Good understanding of the German language
2. Understanding of procedures and risks associated with the study
3. Willing to adhere to the protocol and signing of the consent form
4. Willing to refrain from the consumption of illicit psychoactive substances during the study
5. Willing not to operate heavy machinery within 48 h after administration of a study substance
6. Willing to use effective birth control throughout study participation
7. Body mass index 17 - 34.9 kg/m2

Exclusion Criteria:

1. Relevant chronic or acute medical condition
2. Current or previous major psychiatric disorder (e.g. psychotic disorder)
3. Psychotic disorder or bipolar disorder in first-degree relatives
4. Hypertension (SBP>140/90 mmHg) or hypotension (SBP<85 mmHg)
5. Bradycardia (< 45 bpm)
6. Prolonged QTc interval (males: >450 ms, females: >470 ms)
7. AV block II° (Mobitz type and Webckebach type) and III°
8. Hallucinogenic substance use (not including cannabis) more than 20 times or any time within the previous two months
9. Pregnancy or current breastfeeding
10. Participation in another clinical trial (currently or within the last 30 days)
11. Use of medication that may interfere with the effects of the study medication
12. Tobacco smoking (>10 cigarettes/day)
13. Excessive consumption of alcoholic beverages (>15 drinks/week)

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
1. Altered state of consciousness profile (5D-ASC) | 18 months
  5 Dimensions of Altered States of Consciousness (5D-ASC) consisting of 94 items to be rated on a visual analog scale (0-100 mm), with higher values indicating stronger effects.

SECONDARY OUTCOMES:
Subjective effects (VASs) | 18 months
  Visual Analog Scales assessing the intensity and duration of subjective effects on a scale from 0 - 100 percent with higher scores representing more intense effects.
Mystical-type experiences (PES) | 18 months
  This 100-item Psychedelic Experience Questionnaire/Scale (PES100) is rated on a six-point scale (0 indicating "not at all" and 5 indicatin "extremely"). It comprises distractor items as well as subscales which measure mystical-type effects.
Mystical-type experiences (PAE-PS-ext) | 18 months
  This Phenomenological-Autobiographical-Existential Psychedelic Scale extended (PAE-PS-ext) questionnaire rates psychedelic experiences with a focus on phenomenological, autobiographical, and existential psychedelic experiences (scale from 0 - 100 percent with higher scores representing more intense effects).
3. Emotional breakthrough inventory (EBI+) | 18 months
  This 18-item questionnaire is a visual analog scale (from 0 - 100 percent with higher scores representing more intense effects) assessing emotional breakthrough throughout the study sessions.
Plasma levels of LSD | 18 months
  Assessed 20 times on each study day via blood samples
Plasma levels of psilocybin | 18 months
  Assessed 20 times on each study day via blood samples
Plasma levels of DMT | 18 months
  Assessed 20 times on each study day via blood samples
Plasma levels of ketanserin | 18 months
  Assessed 20 times on each study day via blood samples
Plasma levels of oxytocin | 18 months
  Assessed 2 times on each study day via blood samples
Plasma levels of prolactin | 18 months
  Assessed 2 times on each study day via blood samples
Plasma levels of cortisol | 18 months
  Assessed 2 times on each study day via blood samples
Autonomic effects I | 18 months
  Assessed 16 times on each study day via systolic and diastolic blood pressure
Autonomic effects II | 18 months
  Assessed 16 times on each study day via heart rate
Autonomic effects III | 18 months
  Assessed one time at screening visit and twice on each study day via ECG (QT-time)
Adverse effects (B-LR) | 18 months
  The 2011 revised Beschwerden-Liste (B-LR) consists of a 40-item list covering a wide variety of symptoms and complaints that are answered with a four-point intensity-scoring ranging from 0 indicating "not at all" to 3 indicating "strong."
Adverse effects (SPSI) | 18 months
  The Swiss Psychedelic Side Effects Inventory evaluates side effects associated with psychedelics using a binary "yes or no" approach. Severity is recorded using a three-point intensity scale ranging from 1 indicating "light" to 3 indicating "strong." The impact is recorded using a five-point scale ranging from -2 "very disadvantageous" to +2 "very advantageous." The relation to the drug is recorded using a five-point scale ranging from 0 indicating "unknown" to 4 indicating "certain."
Adverse Events (AE) | 18 months
  Any report of adverse events will be recorded on a AE-Form.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, Prof. Dr. MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital, Basel, Switzerland